CLINICAL TRIAL: NCT05645549
Title: Exploring the Feasibility of Centering Pregnancy With Care Navigation and the Preliminary Effectiveness to Improve Prenatal and Postpartum Appointment Attendance, Maternal and Infant Outcomes, and Access to Social Support Services
Brief Title: Exploring the Feasibility of Centering Pregnancy With Care Navigation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 275134
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centering Pregnancy with Care Navigation for pregnant Marshallese women (Experimental): Forty pregnant Marshallese women will be enrolled in the group prenatal intervention, Centering Pregnancy, with care navigation to determine the feasibility of the intervention and the preliminary effectiveness to improve maternal and infant health care outcomes.
  Interventions: Behavioral: Centering Pregnancy with Care Navigation
- Pregnant Marshallese women enrolled in standard prenatal care (No Intervention): We will use a 1:1 propensity score matching with pregnant Marshallese women who completed standard prenatal care to compare their maternal and infant health care outcomes with those participants enrolled in the intervention.

INTERVENTIONS:
Behavioral: Centering Pregnancy with Care Navigation — Centering Pregnancy is a group based prenatal care intervention. Centering Pregnancy is an evidenced based intervention that has 10 group sessions for pregnant women. Each session has dedicated educational material relative to pregnancy, birth, and infant feeding. In addition, all participants will be provided a bilingual Marshallese care navigator to aid in enrolling them in social support services.
  Arms: Centering Pregnancy with Care Navigation for pregnant Marshallese women

SUMMARY:
Pacific Islanders residing in the United States (US) have disproportionally high rates of preterm birth (<37 weeks) and low birthweight infants (<2,500 grams). They are also more likely to experience preeclampsia, primary cesarean birth, excessive gestational weight gain, and gestational diabetes mellitus (GDM) compared to other racial/ethnic minorities. These maternal health factors serve as precursors to maternal and infant morbidity and mortality. Pacific Islanders have almost twice the infant mortality rate, per 1,000 live births, as compared to non-Hispanic whites and have a higher maternal mortality rate compared to the same group (13.5 verse 12.7). Early and consistent supportive care throughout the pregnancy continuum is strongly associated with positive birth outcomes, including infant and maternal morbidity and mortality, and is a US health priority.

Emerging literature suggests that group-based prenatal programs, like Centering Pregnancy, coupled with care navigation, can mitigate precursors to severe morbidity and mortality. The proposed study will determine the feasibility of Centering Pregnancy with care navigation and the preliminary effectiveness to improve: prenatal and postpartum care appointment attendance, preterm birth, low-birth weight infants, cesarean deliveries, emergency department visits, and access to social support services. Investigators will use a mixed-method approach with two groups of Marshallese participants (propensity score matched on relevant covariates such as maternal age, parity, and sociodemographics), one group in Centering Pregnancy with care navigation and one group from standard prenatal care.

DETAILED DESCRIPTION:
Pacific Islanders residing in the United States (US) have disproportionally high rates of preterm birth (<37 weeks) and low birthweight infants (<2,500 grams). They are also more likely to experience preeclampsia, primary cesarean birth, excessive gestational weight gain, and gestational diabetes mellitus (GDM) compared to other racial/ethnic minorities. These maternal health factors serve as precursors to maternal and infant morbidity and mortality. Pacific Islanders have almost twice the infant mortality rate, per 1,000 live births, as compared to non-Hispanic whites and have a higher maternal mortality rate compared to the same group (13.5 verse 12.7). Early and consistent supportive care throughout the pregnancy continuum is strongly associated with positive birth outcomes, including infant and maternal morbidity and mortality, and is a US health priority.

Emerging literature suggests that group-based prenatal programs, like Centering Pregnancy, coupled with care navigation, can mitigate precursors to severe morbidity and mortality. The proposed study will determine the feasibility of Centering Pregnancy with care navigation and the preliminary effectiveness to improve: prenatal and postpartum care appointment attendance, preterm birth, low-birth weight infants, cesarean deliveries, emergency department visits, and access to social support services. Investigators will use a mixed-method approach with two groups of Marshallese participants (propensity score matched on relevant covariates such as maternal age, parity, and sociodemographics), one group in Centering Pregnancy with care navigation and one group from standard prenatal care. The Specific Aims are:

Aim 1: Determine the feasibility of Centering Pregnancy with care navigation to improve prenatal and postpartum care attendance among Marshallese participants. Hypothesis: Marshallese participants who participate in Centering Pregnancy with care navigation will attend 80% of their prenatal and postpartum care visits.

Aim 2: Determine the preliminary effectiveness of Centering Pregnancy with care navigation to improve maternal health outcomes that can mitigate maternal and infant morbidity and mortality. Hypothesis: Marshallese participants who participate in Centering Pregnancy with care navigation will demonstrate improved maternal health outcomes including: preterm birth, low-birth weight infants, cesarean deliveries, and emergency department visits compared to women receiving standard prenatal care using a propensity score matched comparison group.

Aim 3: Determine the preliminary effectiveness of Centering Pregnancy with care navigation to improve access to social support services to Marshallese participants. Hypothesis: Marshallese particiapnts who have completed Centering Pregnancy with care navigation will report improved access to social support services measured by enrollment in health insurance, maintain insurance post-partum, and access to food, transportation, and housing resources.

ELIGIBILITY:
Inclusion Criteria:

* women who self-report as Marshallese
* 18 years of age or older
* pregnant (12-14 weeks gestation).

Exclusion Criteria:

* conception with the use of fertility treatments
* high-risk pregnancy that requires a transfer to a high-risk clinic
* multiple gestations (i.e. pregnant with more than one infant)
* use of medications known to influence fetal growth (e.g., glucocorticoids, insulin, thyroid, hormones

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with infants that are preterm. | All maternal and infant health records will be collected at six weeks postpartum
  >37 weeks at delivery
Number of participants with infants with low birthweight | All maternal and infant health records will be collected at six weeks postpartum
  <2,500 grams
Number of participants with a caesarean delivery. | All maternal and infant health records will be collected at six weeks postpartum
  the birthing method of infant

SECONDARY OUTCOMES:
The number of social services participants are enrolled in at the end of the intervention. | All social service assessments will take place at six weeks postpartum
  We will assess the enrollment of social services with a bilingual Marshallese care navigator using a mixed methods approach

CONTACTS AND LOCATIONS:
Overall Officials: Britni L Ayers, PhD, Principal Investigator — University of Arkansas for Medical Sciences Northwest
Locations (1):
- University of Arkansas for Medical Sciences-Northwest, Fayetteville, Arkansas, United States